CLINICAL TRIAL: NCT01587404
Title: Relationship Between Catheter Contact Force and Electrogram Characteristics in Fibrillating Human Atrial Myocardium
Brief Title: Catheter Contact Force and Electrograms
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 007856 BLT
Record Dates: First submitted 2012-04-23; First posted 2012-04-30 (Estimated); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Electrogram; Ablation; Contact Force
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Constant Catheter Contact Force (Experimental): No alteration of catheter contact force during recording period
  Interventions: Device: THERMOCOOL® SMARTTOUCH™ Catheter (including Surround Flow)
- Variable catheter contact force (Experimental): change in contact force from low to high after 30seconds of recording.
  Interventions: Device: THERMOCOOL® SMARTTOUCH™ Catheter (including Surround Flow)

INTERVENTIONS:
Device: THERMOCOOL® SMARTTOUCH™ Catheter (including Surround Flow) — Variable contact force as measured at the catheter tip within the left atrium

SUMMARY:
Until recently, there was no way of telling how firmly the tip of the catheter was in contact with the heart and how this contact was orientated. The electrical signals measured through the catheters, known as electrograms, are used to guide the sites and duration of ablation, but the effect of catheter contact and orientation on these signals in human heart muscle that is fibrillating is not known. New catheters have now been developed which can measure the force of contact at their tip: using these, the investigators will examine how contact force affects the electrical behaviour of heart muscle tissue in atrial fibrillation. The effect the force of contact has on the electrogram recorded will also be investigated. In so doing we hope to gain a better understanding of the relationship between tissue contact and the electrograms we measure and in so doing improve the safety and effectiveness of ablation procedures.

Hypothesis: Catheter contact force and orientation have a significant impact on the characteristics of bipolar electrograms in the fibrillating human atrium.

ELIGIBILITY:
Inclusion Criteria:

* Persistent or paroxysmal atrial fibrillation
* Listed for ablation of atrial fibrillation on clinical grounds

Exclusion Criteria:

* Contraindication to catheter ablation
* Contraindication to anticoagulation
* Contraindication to TOE

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2012-04; Primary Completion 2017-05-31 (Actual); Study Completion 2018-08-21 (Actual)

PRIMARY OUTCOMES:
Electrogram characteristics | Baseline and 30 seconds
  Effect of changes in contact force and orientation on: slew rate, local mean cycle length, electrogram complexity and fractionation index, dominant frequency, organisation index, CFAE grade, interval confidence level, shortest complex interval and average complex interval

SECONDARY OUTCOMES:
Electrogram amplitude | Baseline and 30 seconds
Electrogram responses to ablation | Baseline and 30 seconds
  Slew rate, local mean cycle length, electrogram complexity and fractionation index, dominant frequency, organisation index, CFAE grade, interval confidence level, shortest complex interval and average complex interval, amplitude change, AF cycle length, catheter impedance.
Ablation Power (Watts) | Baseline and 30 seconds
  The interaction between catheter contact force and orientation and the power attained during power limited ablation
Electrogram Contact Mapping | During Study
  Use of contact catheters - Constellation and/or PentaRay Catheter to record fibrillatory electrograms and identify areas of interest

CONTACTS AND LOCATIONS:
Overall Officials: Richard J Schilling, MD, Principal Investigator — Professor of Cardiology and Electrophysiology St Barts Hospital and Queen Mary University
Locations (1):
- St Bartholomew's Hospital, London, United Kingdom

REFERENCES:
- [Derived] Ullah W, Hunter RJ, Baker V, Ling LH, Dhinoja MB, Sporton S, Earley MJ, Schilling RJ. Impact of Catheter Contact Force on Human Left Atrial Electrogram Characteristics in Sinus Rhythm and Atrial Fibrillation. Circ Arrhythm Electrophysiol. 2015 Oct;8(5):1030-9. doi: 10.1161/CIRCEP.114.002483. Epub 2015 Jul 7. PMID 26152560
- [Derived] Ullah W, Hunter RJ, Baker V, Dhinoja MB, Sporton S, Earley MJ, Schilling RJ. Target indices for clinical ablation in atrial fibrillation: insights from contact force, electrogram, and biophysical parameter analysis. Circ Arrhythm Electrophysiol. 2014 Feb;7(1):63-8. doi: 10.1161/CIRCEP.113.001137. Epub 2014 Jan 18. PMID 24443504